CLINICAL TRIAL: NCT04362358
Title: Efficacy of an Online Cognitive Behavioral Therapy (CBT) Programme Aiming at Reducing the Stress of Health Workers Involved in the Care of Patients During the Covid-19 Epidemic: a Randomized-controlled Trial
Brief Title: Online Cognitive Behavioral Therapy (CBT) for Stress Disorders in Health Workers Involved in the Care of Patients During the Covid-19 Epidemic
Acronym: REST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7799
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Stress - Prevention of Sleep Disorders, PTSD and Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7 sessions of the online CBT programme (Experimental)
  Interventions: Behavioral: Online cognitive behavioral therapy (CBT)
- Bibliotherapy (Active Comparator)
  Interventions: Behavioral: Online bibliotherapy programme

INTERVENTIONS:
Behavioral: Online cognitive behavioral therapy (CBT) — 7 sessions of Cognitive Behavioural Therapy (CBT) online + possibility to contact the psychological hotline
  Arms: 7 sessions of the online CBT programme
Behavioral: Online bibliotherapy programme — online bibliotherapy programme on the Ma Santé website Also with explanatory sheets and tools to improve stress management and the possibility of contacting the Psychological Hotline
  Arms: Bibliotherapy

SUMMARY:
Some preliminary epidemiological research conduct in China in health workers involved in the care of Covid-19 patients has shown high rates of depression (>50%), generalized anxiety disorder (>44%), insomnia (>36%) and stress symptoms (>73%), which negatively impact their well-being as well as their ability to work effectively . These rates were observed during the epidemic peak, but they can also have a long-term mental health effect, both individually, but also in a systemic manner , similar to what has been reported relative to the SARS-CoV-1 . Cognitive behavioral therapy (CBT) is recognized as an effective treatment for stress-reduction, as well as for the prevention of multiple mental health problems in at-risk individuals . Moreover, CBT has been found to be effective in brief online formats , which could make it feasible during the current Covid-19 epidemic. To our knowledge, there are no online CBT programmes targeting stress problems in health workers involved in the care of patients during the current epidemic context. The aim of our study is to evaluate the efficacy of the online CBT programme we have developped to specifically address immediate perceived stress in health workers, as well as the prevention of mental health problems at 3- and 6-months follow-up

ELIGIBILITY:
Inclusion Criteria:

* Health worker
* Male or Female
* Aged 18-70
* Able to understand the French language

Exclusion Criteria:

* PSS < 16
* Suicidal ideation assessed as < 3 on the item 9 of the PHQ-9
* legally able to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Significant score reduction at the Perceived Stress Scale | T0 inclusion
Significant score reduction at the Perceived Stress Scale | T1 (3-month follow-up)
Significant score reduction at the Perceived Stress Scale | T1 (up to 8 weeks treatment)
Significant score reduction at the Perceived Stress Scale | T2 (6-month follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Weiner, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (1):
- Weiner Luisa, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weiner L, Berna F, Nourry N, Severac F, Vidailhet P, Mengin AC. Efficacy of an online cognitive behavioral therapy program developed for healthcare workers during the COVID-19 pandemic: the REduction of STress (REST) study protocol for a randomized controlled trial. Trials. 2020 Oct 21;21(1):870. doi: 10.1186/s13063-020-04772-7. PMID 33087178